CLINICAL TRIAL: NCT01899963
Title: Time to Treatment Utilizing a Tele-Retinal Referral System for Wet Age Related Macular Degeneration and Diabetic Macular Edema: A Pilot Study
Brief Title: Time to Treatment Utilizing a Tele-Retinal Referral System for wAMD and DME: A Pilot Study
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Other Study IDs: Tele-retinal Referral T.T.T.
Record Dates: First submitted 2013-07-09; First posted 2013-07-16 (Estimated); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Wet Age Related Macular Degeneration; Diabetic Macular Edema
Keywords: wet Age Related Macular Degeneration; Diabetic Macular Edema; Telemedicine; Teleophthalmology; Time to Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Tele-ophthalmology Referral Group: This group includes patients referred to a retinal specialist via a teleophthalmology referral system.
- Conventional Referral Group: This group includes patients referred to a retinal specialist via a conventional fax system.

SUMMARY:
In this province, optometrists are often responsible for contacting the retinal specialists' office to arrange patients to be examined for suspected emergencies or more routine referrals related to the eye. This is often done by faxing a referral form to the specialists' office, where the retinal specialist will examine the information presented in the referral form and make a decision on when the patient should be seen. This current method has some important considerations, such as the difficulty of transmitting clear images of the back of the eye over fax. Having this information could help the retinal specialist in determining when the patient should be seen, especially in terms of booking additional tests or when treatment should be given.

Teleophthalmology is a branch of telemedicine that delivers eye care through digital equipment and telecommunications technology. It offers some unique advantages, such as the ability to be integrated with electronic health records, the ability to be viewed by multiple members of the health care team, and potentially reduce wait times and travel times to the ophthalmologist.

However, there is no comparison known to the study team between whether patients being referred from optometrists to retina specialists through a teleophthalmology system will be treated earlier than patients through a conventional fax system. This study aims to examine and provide more information on this topic.

DETAILED DESCRIPTION:
Within the province of Ontario, there are a limited number of retinal specialists for a large and geographically diverse population of 13.5 million people in 2012. Because the majority of these specialists are located in larger urban centers, many rural patients have difficulty travelling the significant distance from their communities to the city. Currently in Ontario optometrists are responsible for triaging retinal eye diseases; emergency referrals such as endophthalmitis are organized by same-day telephone consultations, while more routine referrals are scheduled by fax.

This current method of triage has particular important considerations. Because of the limited number of retinal specialists long wait times can lead to permanent vision loss if the referral is inaccurate, where the patient should have been seen and treated sooner instead of later such as the case of wet age-related macular degeneration (wAMD) and Diabetic Macular Edema (DME). In addition, essential vision tests such as fluorescein angiography (FA) are often available only in a hospital setting rather within physician or optometrists' office. For patients from rural or remote communities, this inconvenience could result in lost wages, a long return trip back the next day or even an overnight stay.

Teleophthalmology is a branch of telemedicine that delivers eye care through digital equipment and telecommunications technology. It offers some unique advantages, such as the ability to be integrated with electronic health records, the ability to be viewed by multiple members of the health care team, and potentially reduce wait times and travel times to the ophthalmologist. Within Canada, there have been different teleophthalmology initiatives to provide access to specialists to optometrists and primary care practitioners particularly in rural and remote areas, improving ophthalmologic care and reducing unnecessary patient travel expenditures. These teleophthalmology systems can include fundus and Optical Coherence Tomography (OCT) images to aid the ophthalmologist in more accurately diagnosing and triaging the referral. Hanson et al. in a retrospective case series noted that tele-referrals to retinal specialists from optometrists reduced average travel time, travel distance and the number of office visits to retina specialists while improving efficiency of clinical examination, testing, and treatment.

However, there currently is no research known to the study team that actively compares the time to treatment for patients based on teleophthalmology referral and assessment versus a conventional paper referral system from optometrists to retinal specialists. For conditions like wAMD and DME related to Diabetic Retinopathy that are often referred via teleophthalmology, the difference in time to treatment could prevent vision loss. The inclusion of fundus and OCT images in teleophthalmology could also improve triage accuracy and prioritization of referrals and appointments to the retinal specialist. This study focuses on comparing the time to treatment for a tele-retinal referral system to a paper referral system by focusing on two prevalent retinal conditions: wet AMD and DME. The results could demonstrate that tele-ophthalmology can reduce the time to treatment for patients with wet AMD and DME in Ontario, improving access to retinal specialists and allowing for more efficient triage of patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged greater than 18 years,
* Able to provide informed consent,
* Referred from an optometrist either participating in the teleophthalmology referral system or via conventional fax referrals with a provisional diagnosis of possible wet AMD or DME to any of the physician investigators.

Exclusion Criteria:

* Patients with a presumed diagnosis of wet AMD and/or DME at the time of referral who previously had diagnostic imaging (ex. fundus images, OCT images) performed as part of the referral will be excluded;
* Patients unable to tolerate fluorescein angiography (FA);
* Patients unable to travel to the retina practice for treatment or further testing,
* Patients unable to fully understand the study requirements and provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients who are referred from an optometrist either participating in the teleophthalmology referral system or via conventional fax referrals with a provisional diagnosis of possible wet AMD or DME to any of the physician investigators.
Sampling Method: Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2022-01 (Actual); Study Completion 2022-02 (Actual)

PRIMARY OUTCOMES:
Time to Treatment | Average 5-6 Weeks.
  Defined as defined as the time between when the retina specialist reviews the information collected by either system to when the patient receives treatment by the specialist in the clinic.

SECONDARY OUTCOMES:
Maximum wait time | Can range from 2-6 weeks.
  Maximum time between assessment and further assessment, testing, or treatment.
Minimum Wait Time | Can range from 2-6 weeks.
  Minimum time between assessment and further assessment, testing, or treatment for patients in either cohort.
Mean wait time | Can range from 2-6 weeks.
  Mean time between patients of a single cohort for further assessment, testing, or treatment.
Travel time | Can range from 30 minutes or greater.
  This will serve to examine if there is a decreased frequency of visits and subsequently reduced travel time for office visits, for assessment, treatment, or testing for the ophthalmology referral group compared to the fax referral group.
Travel Distance | Can range from 1 kilometer or greater.
  This will serve to examine if there is a decreased frequency of travel in terms of distance for office visits for assessment, treatment, or testing for the ophthalmology referral group compared to the fax referral group.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Healthcare Hamilton King Campus, Hamilton, Ontario, Canada